CLINICAL TRIAL: NCT05141539
Title: Rehabilitation Assessment and Progress Tracking System Based on Video Images for Dysphagic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: COA. MURA2021/73
Record Dates: First submitted 2021-11-25; First posted 2021-12-02 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Healthy; Head and Neck Cancer
Keywords: Head and Neck Neoplasms; DNA Damage; Fibrosis; Humans Inflammation; Neoplasms; Radiation Injuries; Radiotherapy; Transforming Growth Factor beta
MeSH Terms: conditions — Head and Neck Neoplasms; Fibrosis; Neoplasms; Radiation Injuries; Camurati-Engelmann Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation assessment software (Experimental): This arm applies the developed rehabilitation assessment software by using two web cameras placed in the front and the side of the subject. The subject sits between two cameras. The observer asks the subject to move the head in each direction, to open the mouth, and to move the tongue. The software will measure CROM, mouth opening, and tongue movement.
  Interventions: Device: Rehabilitation assessment software
- video-fluoroscopic swallowing and FOIS. (Experimental): This arm applies video-fluoroscopic swallowing (VFSS) and functional oral intake scale (FOIS) to measure the direct, dynamic view of oral, pharyngeal, and upper esophageal function during swallowing with food and liquid mixed with barium, and the functional intake of dysphagic patients, respectively.
  Interventions: Device: Rehabilitation assessment software; Device: VFSS and FOIS

INTERVENTIONS:
Device: Rehabilitation assessment software — In phase 2, this software will be tested in occupational therapists, and head and neck cancer patients results for reliability and validity.
  In phase 3, the experiment in the oropharyngeal dysphagia specialists results in content validity, the comparison between the developed software, and VFSS and FOIS results in criterion-related validity, and the experiment in head and neck cancer patients results in reliability.
Device: VFSS and FOIS — In phase 3, this study applies VFSS and FOIS for the head and neck cancer patients for comparison with the developed rehabilitation assessment software for criterion-related validity.
  Arms: video-fluoroscopic swallowing and FOIS.

SUMMARY:
The current cervical range of motion (CROM) and tongue movement measurement methods are not reliable between observers, which is not practical in real-world usage. This research is to develop the cervical range of motion measurement, and tongue movement estimation software, to compare between the developed software and the current measurement techniques, and to test in clinical aspects for reliability and validity assessment. The investigators investigate the developed software in healthy people in phase 1. In phases 2 and 3, the investigators compare the software to the standard measurement methods in dysphagic patients who have head and neck cancer for reliability and validity.

ELIGIBILITY:
Inclusion Criteria in Phase 2

* Occupational therapist

  1. This study requires the subject to be between 18 and 80 years old.
  2. The subject needs to be Thai.
  3. The subject can communicate in the Thai language.
  4. Working as an occupational therapist in Ramathibodhi hospital.
  5. The subject is consent.
* Head and neck cancer patients

  1. This study requires the subject to be between 18 and 80 years old.
  2. The subject needs to have stable vital signs.
  3. The subject can make the body steady sit on the chair longer than 30 minutes.
  4. The subject is diagnosed with head and neck cancer and treated at Ramathibodhi hospital.
  5. Eating Assessment Tool (EAT-10) score is more than or equals 3.
  6. Montreal Cognitive Assessment (MOCA) score is more than or equals 23.
  7. The subject is consent.

Exclusion Criteria in Phase 2

* Occupational therapist

  1. Cannot participate in the experiment.
  2. The therapist denied or withdrew.
* Head and neck cancer patients

  1. Have pain around the examination area such as oral mucosa, tongue, and neck.
  2. Participate in chemotherapy.
  3. Cannot participant until the end of the experiment.
  4. The subject denied or withdrew.

Inclusion Criteria in Phase 3

* Dysphagic Specialist

  1. The age is more than 18 years old.
  2. The specialist is required to be Thai.
  3. The specialist can communicate in the Thai language.
  4. Working in oropharyngeal swallowing rehabilitation in the dysphagic unit at Ramathibodhi hospital for more than 3 years.
  5. The specialist has papers related to swallowing rehabilitation.
  6. The specialist is consent.
* Observers

  1. This study requires the subject to be between 18 and 80 years old.
  2. The observer can communicate in the Thai language.
  3. The observer needs to be Thai.
  4. Working in swallowing rehabilitation in Ramathibodhi hospital for more than a year.
  5. The observer is consent.
* Head and neck cancer patients The criteria are the same as the inclusion criteria of head and neck cancer patients in phase 2.

Exclusion Criteria in Phase 3

* Dysphagic Specialist

  1. Cannot participant in the experiment.
  2. The specialist denied or withdrew.
* Observers

  1. Have a relationship with software development.
  2. Cannot participate in the study until the end of the experiment.
  3. The subject denied or withdrew.
* Head and neck cancer patients The criteria are the same as the exclusion criteria of head and neck cancer patients in phase 2.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Intra-rater reliability between the developed rehabilitation assessment software and the standard CROM measurement method. | One hour
  The same investigator will repeat cervical range of motion measurement by using the developed rehabilitation software and the standard cervical range of motion (CROM) measurement method from the goniometer.
Inter-rater reliability between the developed rehabilitation assessment software and the standard CROM measurement method. | One hour
  The cervical range of motion (CROM) measurement by using the developed rehabilitation software and the standard CROM measurement method from the goniometer will be repeated by different observers.
Concurrent measurement validity between the developed rehabilitation assessment software and the standard CROM measurement method. | One hour
  The correlation of the concurrent cervical range of motion (CROM) measurement outcome at approximately the same time between the developed rehabilitation assessment software and the standard CROM measurement method from the goniometer.
Criterion-related validity between the developed rehabilitation assessment software, and VFSS and FOIS. | One month
  The criterion-related validity of the rehabilitation assessment software will be assessed by the correlation between the cervical range of motion measurement by the developed rehabilitation assessment software and the functional swallowing assessment by videofluoroscopic Swallowing Study (VFSS), and functional oral intake scale (FOIS).

CONTACTS AND LOCATIONS:
Overall Officials: Panrasee Ritthipravat, Principal Investigator — Mahidol University
Locations (1):
- Department of Rehabilitation Medicine, Ramathibodhi Hospital, Phaya Thai, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
The data requires to be confidential. It is prohibited to share the participant-level data.